CLINICAL TRIAL: NCT01054729
Title: A Multi-center, Double-Blind, Parallel Group, Randomized, Placebo-Controlled, Dose Ranging Study to Investigate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics Following Oral Administration of PSI-7977 in Combination With Standard of Care (Pegylated Interferon and Ribavirin) in Treatment-Naïve Patients With Chronic HCV Infection Genotype 1
Brief Title: Dose-Ranging Study of Sofosbuvir in Combination With Pegylated Interferon and Ribavirin in Treatment Naïve GT 1 HCV Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: P7977-0221
Record Dates: First submitted 2010-01-21; First posted 2010-01-22 (Estimated); Results first posted 2014-02-19 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2014-03

CONDITIONS: Hepatitis C
Keywords: Chronic Hepatitis C infection Genotype 1; HCV; GT1; GT 1
MeSH Terms: conditions — Hepatitis C | interventions — Sofosbuvir; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sofosbuvir 100 mg+PEG+RBV (Experimental): Participants received sofosbuvir 100 mg (1 x 100 mg tablet) and placebo to match sofosbuvir (3 tablets) for 28 days (baseline to Day 28), plus PEG+RBV (baseline to Week 48)
  Interventions: Drug: Sofosbuvir; Drug: PEG; Drug: RBV
- Sofosbuvir 200 mg+PEG+RBV (Experimental): Participants received sofosbuvir 200 mg (2 x 100 mg tablets) and placebo to match sofosbuvir (2 tablets) for 28 days (baseline to Day 28), plus PEG+RBV (baseline to Week 48)
  Interventions: Drug: Sofosbuvir; Drug: PEG; Drug: RBV
- Sofosbuvir 400 mg+PEG+RBV (Experimental): Participants received sofosbuvir 400 mg (4 x 100 mg tablets) for 28 days (baseline to Day 28), plus PEG+RBV (baseline to Week 48)
  Interventions: Drug: Sofosbuvir; Drug: PEG; Drug: RBV
- Placebo+PEG+RBV (Active Comparator): Participants received placebo to match sofosbuvir (4 tablets) for 28 days (baseline to Day 28), plus PEG+RBV (baseline to Week 48)
  Interventions: Drug: Placebo; Drug: PEG; Drug: RBV

INTERVENTIONS:
Drug: Sofosbuvir — Sofosbuvir tablet(s) administered orally once daily
  Other Names: Sovaldi®; GS-7977; PSI-7977
  Arms: Sofosbuvir 100 mg+PEG+RBV; Sofosbuvir 200 mg+PEG+RBV; Sofosbuvir 400 mg+PEG+RBV
Drug: Placebo — Placebo to match sofosbuvir administered orally once daily
  Arms: Placebo+PEG+RBV
Drug: PEG — Pegylated interferon alfa-2a (PEG) 180 μg was administered once weekly by subcutaneous injection.
  Other Names: Pegasys®
Drug: RBV — Ribavirin (RBV) tablets were administered orally in a divided daily dose according to package insert weight-based dosing recommendations (< 75kg = 1000 mg and ≥ 75 kg = 1200 mg).
  Other Names: Copegus®

SUMMARY:
Participants with genotype 1 HCV infection were randomized to 1 of 3 sofosbuvir doses (100 mg, 200 mg, or 400 mg) or matching placebo once daily based upon stratification for IL28B status (CC or CT/TT). Placebo tablets were administered to participants receiving 100 mg active sofosbuvir (3 placebo tablets) and 200 mg active sofosbuvir (2 placebo tablets) in order to maintain the study blind. Participants received sofosbuvir/matching placebo from Day 0 to 27. Participants also received treatment with PEG+RBV starting on Day 0 of the study which continued for 48 weeks. Participants were evaluated for sustained virologic response (SVR) for an additional 24 weeks following completion of study treatment.

ELIGIBILITY:
Inclusion Criteria:

* Treatment-naive males and females, 18-65 years of age
* Genotype 1 HCV infection
* Negative pregnancy test for females of childbearing age
* Females of childbearing age and males with female partners of childbearing age must use two forms of contraception during treatment and following the last dose of ribavirin in accordance with locally approved label for ribavirin

Exclusion Criteria:

* Hepatitis B or HIV infection
* Pregnant or breast feeding females or male partners of pregnant females
* Previous interferon or ribavirin-based therapy or investigational anti-HCV agent
* History or evidence of medical condition associated with chronic liver disease other than HCV

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2010-01; Primary Completion 2010-04 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert H. Hyland, DPhil, Study Director — Gilead Sciences
Locations (7):
- United States (6):
  - Quest Clinical Research, San Francisco, California
  - University of Florida, Gainesville, Florida
  - Orlando Immunology Center, Orlando, Florida
  - Duke University, Durham, North Carolina
  - Alamo Medical Research Center, San Antonio, Texas
  - Virginia Mason Medical Center, Seattle, Washington
- Fundacion de Investigacion de Diego, Santurce, Puerto Rico, Puerto Rico

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at a total of 7 study sites in the United States. The first participant was screened on 18 January 2010. The last participant observation was on 25 August 2011.
Pre-assignment Details: 143 participants were screened and 64 were randomized; 63 participants were treated, and comprise the Safety Analysis Set.
Groups:
- Sofosbuvir 100 mg+PEG+RBV: Participants received sofosbuvir 100 mg for 28 days (baseline to Day 28), plus PEG+RBV (baseline to Week 48)
- Sofosbuvir 200 mg+PEG+RBV: Participants received sofosbuvir 200 mg for 28 days (baseline to Day 28), plus PEG+RBV (baseline to Week 48)
- Sofosbuvir 400 mg+PEG+RBV: Participants received sofosbuvir 400 mg for 28 days (baseline to Day 28), plus PEG+RBV (baseline to Week 48)
- Placebo+PEG+RBV: Participants received placebo to match sofosbuvir for 28 days (baseline to Day 28), plus PEG+RBV (baseline to Week 48)
Period: Overall Study
Arm/Group | Sofosbuvir 100 mg+PEG+RBV | Sofosbuvir 200 mg+PEG+RBV | Sofosbuvir 400 mg+PEG+RBV | Placebo+PEG+RBV
Started | 16 | 19 | 15 | 14
Randomized and Treated | 16 | 18 | 15 | 14
Completed | 12 | 14 | 9 | 11
Not Completed | 4 | 5 | 6 | 3
Not completed — Randomized but Not Treated | 0 | 1 | 0 | 0
Not completed — Adverse Event | 1 | 1 | 2 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up, Later Contacted Site | 0 | 1 | 0 | 0
Not completed — Non-responder | 1 | 0 | 1 | 1
Not completed — PEG/RBV Non-responder | 1 | 0 | 1 | 0
Not completed — Personal/Obligations | 0 | 1 | 0 | 0
Not completed — Subject moved | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participants who were randomized and treated were analyzed for Baseline Characteristics
Groups:
- Sofosbuvir 100 mg+PEG+RBV: Sofosbuvir 100 mg for 28 days plus PEG+RBV for 48 weeks
- Sofosbuvir 200 mg+PEG+RBV: Sofosbuvir 200 mg for 28 days plus PEG+RBV for 48 weeks
- Sofosbuvir 400 mg+PEG+RBV: Sofosbuvir 400 mg for 28 days plus PEG+RBV for 48 weeks
- Placebo+PEG+RBV: Placebo to match sofosbuvir for 28 days plus PEG+RBV for 48 weeks
- Total: Total of all reporting groups
Arm/Group | Sofosbuvir 100 mg+PEG+RBV | Sofosbuvir 200 mg+PEG+RBV | Sofosbuvir 400 mg+PEG+RBV | Placebo+PEG+RBV | Total
Number analyzed (Participants) | 16 | 18 | 15 | 14 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.4 (10.10) | 44.4 (8.34) | 44.9 (8.43) | 46.6 (11.44) | 45.0 (9.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 4 | 3 | 20
  Male | 11 | 10 | 11 | 11 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 9 | 8 | 4 | 28
  Not Hispanic or Latino | 9 | 9 | 7 | 10 | 35
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska native | 0 | 0 | 1 | 0 | 1
  Black or African American | 1 | 2 | 2 | 0 | 5
  White | 15 | 16 | 12 | 14 | 57
Hepatitis C (HCV) RNA [Mean (Standard Deviation); unit: log10 IU/mL] | 6.64 (0.476) | 6.28 (0.813) | 6.49 (0.602) | 6.48 (0.666) | 6.47 (0.655)
HCV RNA Level (IU/mL) [Number; unit: participants]
  ≤ 800,000 | 1 | 3 | 3 | 4 | 11
  > 800,000 | 15 | 15 | 12 | 10 | 52
Liver Biopsy Fibrosis Score [Number; unit: participants]
  None or Minimal Fibrosis | 5 | 6 | 5 | 4 | 20
  Portal Fibrosis | 11 | 10 | 9 | 9 | 39
  Bridging Fibrosis | 0 | 2 | 1 | 1 | 4
  Cirrhosis | 0 | 0 | 0 | 0 | 0
Alanine Aminotransferase (ALT) [Mean (Standard Deviation); unit: IU/L] | 69.0 (29.69) | 72.6 (46.45) | 95.4 (75.86) | 70.0 (40.73) | 76.2 (50.08)
IL28b Genotype [Number; unit: participants] — CC, CT, and TT alleles are different forms of the IL28b gene.
  participants
    CC | 4 | 5 | 4 | 4 | 17
    CT/TT | 12 | 13 | 11 | 10 | 46

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experienced Adverse Events During the Sofosbuvir Treatment Period
Description: Adverse events (AEs) occurring during the sofosbuvir treatment period were summarized across the participant population. A participant was counted once if they had a qualifying event.
Time Frame: Baseline to Week 4
Population: Safety Analysis Set: participants were randomized and received at least 1 dose of study drug
Measure: Number; unit: percentage of participants
Arm/Group | Sofosbuvir 100 mg+PEG+RBV | Sofosbuvir 200 mg+PEG+RBV | Sofosbuvir 400 mg+PEG+RBV | Placebo+PEG+RBV
Number analyzed (Participants) | 16 | 18 | 15 | 14
percentage of participants
  Any AE | 87.5 | 83.3 | 86.7 | 85.7
  Drug-related AE | 12.5 | 27.8 | 33.3 | 42.9
  Grade 3 or higher AE | 0.0 | 0.0 | 0.0 | 0.0
  AE leading to drug discontinuation/interruption | 0.0 | 0.0 | 0.0 | 0.0
  Serious AE | 0.0 | 0.0 | 0.0 | 0.0

2. Secondary Outcome: Change in Circulating HCV RNA at Week 4
Time Frame: Baseline to Week 4
Population: Safety Analysis Set
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Sofosbuvir 100 mg+PEG+RBV | Sofosbuvir 200 mg+PEG+RBV | Sofosbuvir 400 mg+PEG+RBV | Placebo+PEG+RBV
Number analyzed (Participants) | 16 | 18 | 15 | 14
log10 IU/mL | -5.323 (0.6642) | -5.081 (0.8068) | -5.346 (0.6130) | -2.8 (1.6034)

3. Secondary Outcome: Percentage of Participants With Rapid Virologic Response at Week 4
Description: Rapid virologic response (RVR) was defined as HCV RNA below the limit of detection (LOD [15 IU/mL]) at Week 4.
Time Frame: Week 4
Population: Safety Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Sofosbuvir 100 mg+PEG+RBV | Sofosbuvir 200 mg+PEG+RBV | Sofosbuvir 400 mg+PEG+RBV | Placebo+PEG+RBV
Number analyzed (Participants) | 16 | 18 | 15 | 14
percentage of participants | 87.5 | 94.4 | 93.3 | 21.4

4. Secondary Outcome: Percentage of Participants With Sustained Virologic Response (SVR) at 12 and 24 Weeks After Last Dose of PEG+RBV Following Completion of 48 Weeks of Treatment
Description: SVR at 12 weeks (SVR12) and 24 weeks (SVR24) was defined as HCV RNA < LOD 12 and 24 weeks after last dose of PEG+RBV, respectively, following completion of 48 weeks of treatment (4 weeks of sofosbuvir or matching placebo and PEG+RBV, followed by an additional 44 weeks of PEG+RBV).
Time Frame: Post-treatment Weeks 12 and 24
Population: Safety Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Sofosbuvir 100 mg+PEG+RBV | Sofosbuvir 200 mg+PEG+RBV | Sofosbuvir 400 mg+PEG+RBV | Placebo+PEG+RBV
Number analyzed (Participants) | 16 | 18 | 15 | 14
percentage of participants
  SVR12 | 56.3 | 72.2 | 86.7 | 50.0
  SVR24 | 56.3 | 83.3 | 80.0 | 42.9

5. Secondary Outcome: Plasma Pharmacokinetics of Sofosbuvir: Cmax at Day 0
Description: The Cmax of sofosbuvir was measured at Day 0 following a single dose of sofosbuvir.
  Cmax is defined as the maximum concentration of drug.
Time Frame: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 12 hours postdose
Population: Participants in the Safety Analysis Set with available data and who received a regimen containing sofosbuvir were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sofosbuvir 100 mg+PEG+RBV | Sofosbuvir 200 mg+PEG+RBV | Sofosbuvir 400 mg+PEG+RBV
Number analyzed (Participants) | 16 | 17 | 15
ng/mL | 218.08 (181.54) | 332.26 (215.53) | 1257.50 (736.36)

6. Secondary Outcome: Plasma Pharmacokinetics of Sofosbuvir: Cmax at Day 27
Description: The Cmax of sofosbuvir was measured at Day 27 following continuous dosing of sofosbuvir.
Time Frame: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 24 hours postdose)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sofosbuvir 100 mg+PEG+RBV | Sofosbuvir 200 mg+PEG+RBV | Sofosbuvir 400 mg+PEG+RBV
Number analyzed (Participants) | 16 | 16 | 15
ng/mL | 253.54 (171.10) | 475.14 (358.88) | 1355.65 (853.85)

7. Secondary Outcome: Plasma Pharmacokinetics of Sofosbuvir: AUCinf at Day 0
Description: The AUCinf of sofosbuvir was analyzed at Day 0 (following a single dose of sofosbuvir).
  AUCinf is defined as the concentration of drug (area under the plasma concentration versus time curve) extrapolated to infinite time.
Time Frame: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 12 hours postdose
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Sofosbuvir 100 mg+PEG+RBV | Sofosbuvir 200 mg+PEG+RBV | Sofosbuvir 400 mg+PEG+RBV
Number analyzed (Participants) | 16 | 17 | 15
h*ng/mL | 280.19 (199.54) | 585.56 (342.53) | 1867.24 (959.30)

8. Secondary Outcome: Plasma Pharmacokinetics of Sofosbuvir: AUCtau at Day 27
Description: The AUCtau of sofosbuvir was analyzed at Day 27 (following continuous dosing of sofosbuvir).
  AUCtau is defined as the concentration of drug (area under the plasma concentration versus time curve) over the dosing interval.
Time Frame: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 24 hours postdose)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Sofosbuvir 100 mg+PEG+RBV | Sofosbuvir 200 mg+PEG+RBV | Sofosbuvir 400 mg+PEG+RBV
Number analyzed (Participants) | 16 | 16 | 15
h*ng/mL | 375.70 (203.13) | 732.27 (297.19) | 2011.23 (988.25)

9. Secondary Outcome: Plasma Pharmacokinetics of GS-331007: Cmax at Day 0
Description: The Cmax of GS-331007 was measured at Day 0 following a single dose of sofosbuvir. GS-331007 is the predominant circulating metabolite of sofosbuvir.
Time Frame: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 12 hours postdose
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sofosbuvir 100 mg+PEG+RBV | Sofosbuvir 200 mg+PEG+RBV | Sofosbuvir 400 mg+PEG+RBV
Number analyzed (Participants) | 16 | 17 | 15
ng/mL | 197.32 (88.68) | 357.33 (99.88) | 662.13 (214.76)

10. Secondary Outcome: Plasma Pharmacokinetics of GS-331007: Cmax at Day 27
Description: The Cmax of GS-331007 was measured at Day 27 following continuous dosing of sofosbuvir.
Time Frame: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 24 hours postdose)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sofosbuvir 100 mg+PEG+RBV | Sofosbuvir 200 mg+PEG+RBV | Sofosbuvir 400 mg+PEG+RBV
Number analyzed (Participants) | 16 | 16 | 15
ng/mL | 233.79 (105.02) | 357.38 (109.91) | 717.23 (208.62)

11. Secondary Outcome: Plasma Pharmacokinetics of GS-331007: AUCinf at Day 0
Description: The AUCinf of GS-331007 was analyzed at Day 0 (following a single dose of sofosbuvir).
Time Frame: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 12 hours postdose
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Sofosbuvir 100 mg+PEG+RBV | Sofosbuvir 200 mg+PEG+RBV | Sofosbuvir 400 mg+PEG+RBV
Number analyzed (Participants) | 16 | 17 | 15
h*ng/mL | 2173.18 (852.32) | 3984.88 (895.69) | 7559.91 (3065.23)

12. Secondary Outcome: Plasma Pharmacokinetics of GS-331007: AUCtau at Day 27
Description: The AUCtau of GS-331007 was analyzed at Day 27 (following continuous dosing of sofosbuvir).
Time Frame: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 24 hours postdose)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Sofosbuvir 100 mg+PEG+RBV | Sofosbuvir 200 mg+PEG+RBV | Sofosbuvir 400 mg+PEG+RBV
Number analyzed (Participants) | 16 | 16 | 15
h*ng/mL | 2256.81 (982.40) | 3389.23 (832.01) | 7398.99 (2633.70)

13. Secondary Outcome: Plasma Pharmacokinetics of GS-566500: Cmax at Day 0
Description: The Cmax of GS-566500 was measured at Day 0 following a single dose of sofosbuvir. GS-566500 is one of the major metabolites of sofosbuvir.
Time Frame: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 12 hours postdose
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sofosbuvir 100 mg+PEG+RBV | Sofosbuvir 200 mg+PEG+RBV | Sofosbuvir 400 mg+PEG+RBV
Number analyzed (Participants) | 16 | 17 | 15
ng/mL | 69.99 (35.98) | 145.51 (31.95) | 293.35 (92.75)

14. Secondary Outcome: Plasma Pharmacokinetics of GS-566500: Cmax at Day 27
Description: The Cmax of GS-566500 was measured at Day 27 following continuous dosing of sofosbuvir.
Time Frame: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 24 hours postdose)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sofosbuvir 100 mg+PEG+RBV | Sofosbuvir 200 mg+PEG+RBV | Sofosbuvir 400 mg+PEG+RBV
Number analyzed (Participants) | 16 | 16 | 15
ng/mL | 64.75 (38.51) | 132.72 (49.33) | 237.46 (51.66)

15. Secondary Outcome: Plasma Pharmacokinetics of GS-566500: AUCinf at Day 0
Description: The AUCinf of GS-566500 was analyzed at Day 0 (following a single dose of sofosbuvir).
Time Frame: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, and 12 hours postdose
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Sofosbuvir 100 mg+PEG+RBV | Sofosbuvir 200 mg+PEG+RBV | Sofosbuvir 400 mg+PEG+RBV
Number analyzed (Participants) | 16 | 17 | 15
h*ng/mL | 266.22 (122.40) | 645.95 (228.09) | 1315.94 (618.96)

16. Secondary Outcome: Plasma Pharmacokinetics of GS-566500: AUCtau at Day 27
Description: The AUCtau of GS-566500 was analyzed at Day 27 (following continuous dosing of sofosbuvir).
Time Frame: Predose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, and 24 hours postdose)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Sofosbuvir 100 mg+PEG+RBV | Sofosbuvir 200 mg+PEG+RBV | Sofosbuvir 400 mg+PEG+RBV
Number analyzed (Participants) | 16 | 16 | 15
h*ng/mL | 262.00 (120.64) | 571.95 (156.59) | 1072.91 (327.09)

17. Secondary Outcome: Percentage of Participants Who Developed Resistance to Sofosbuvir
Time Frame: Baseline to Week 4
Population: Participants in the Safety Analysis Set who received a regimen containing sofosbuvir were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Sofosbuvir 100 mg+PEG+RBV | Sofosbuvir 200 mg+PEG+RBV | Sofosbuvir 400 mg+PEG+RBV
Number analyzed (Participants) | 16 | 18 | 15
percentage of participants | 0.0 | 0.0 | 0.0

ADVERSE EVENTS:
Time Frame: Baseline to Week 48
Arm/Group | Sofosbuvir 100 mg+PEG+RBV | Sofosbuvir 200 mg+PEG+RBV | Sofosbuvir 400 mg+PEG+RBV | Placebo+PEG+RBV
Serious Adverse Events (participants affected / at risk) | 1/16 | 0/18 | 3/15 | 1/14
Other Adverse Events (participants affected / at risk) | 14/16 | 18/18 | 13/15 | 13/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sofosbuvir 100 mg+PEG+RBV (N=16) | Sofosbuvir 200 mg+PEG+RBV (N=18) | Sofosbuvir 400 mg+PEG+RBV (N=15) | Placebo+PEG+RBV (N=14)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sofosbuvir 100 mg+PEG+RBV (N=16) | Sofosbuvir 200 mg+PEG+RBV (N=18) | Sofosbuvir 400 mg+PEG+RBV (N=15) | Placebo+PEG+RBV (N=14)
Anaemia (Blood and lymphatic system disorders) | 0 | 8 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 3 | 0 | 1
Motion sickness (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Blepharitis (Eye disorders) | 1 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 1
Eye pain (Eye disorders) | 0 | 0 | 1 | 0
Presbyopia (Eye disorders) | 0 | 0 | 0 | 1
Retinal vasculitis (Eye disorders) | 0 | 0 | 1 | 0
Retinitis (Eye disorders) | 1 | 0 | 0 | 0
Visual acuity reduced (Eye disorders) | 1 | 1 | 2 | 1
Visual impairment (Eye disorders) | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 2 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 5 | 6 | 9 | 6
Retching (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 3 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0
Chills (General disorders) | 7 | 6 | 4 | 2
Fatigue (General disorders) | 7 | 8 | 9 | 8
Injection site erythema (General disorders) | 1 | 2 | 0 | 1
Injection site irritation (General disorders) | 0 | 1 | 0 | 0
Injection site reaction (General disorders) | 1 | 1 | 1 | 2
Irritability (General disorders) | 1 | 0 | 1 | 2
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1
Pain (General disorders) | 1 | 2 | 1 | 3
Pyrexia (General disorders) | 2 | 1 | 1 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0 | 1
Impetigo (Infections and infestations) | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Weight increased (Investigations) | 0 | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 1 | 3 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 2 | 3 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 1 | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Balance disorder (Nervous system disorders) | 1 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 1 | 3 | 2
Headache (Nervous system disorders) | 4 | 6 | 5 | 2
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0
Sinus headache (Nervous system disorders) | 0 | 1 | 0 | 0
Affect lability (Psychiatric disorders) | 1 | 2 | 1 | 2
Anxiety (Psychiatric disorders) | 2 | 1 | 3 | 0
Daydreaming (Psychiatric disorders) | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 2 | 2 | 0
Insomnia (Psychiatric disorders) | 5 | 3 | 3 | 2
Mood swings (Psychiatric disorders) | 0 | 1 | 1 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Sexual dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 3 | 2 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 3 | 5 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 2
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Flushing (Vascular disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years